CLINICAL TRIAL: NCT01956188
Title: Efficacy of EPA and DHA Supplementation in Systemic Lupus Erythematosus and Primary Antiphospholipid Syndrome
Brief Title: Omega 3 in LES and APS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fabiana Braga Benatti, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Omega 3 and SLE and APS USP
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Systemic Lupus Erythematosus; Primary Antiphospholipid Syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPA and DHA supplementation (Experimental): EPA (1800mg/d) and DHA (1200mg/d) supplementation
  Interventions: Dietary Supplement: EPA and DHA supplementation
- Placebo (Placebo Comparator): Soy oil (3000 mg/d)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EPA and DHA supplementation — Subjects will be given 3g/d (1,2g of DHA and 1,8g of EPA) - 5 capsules per day.
  Arms: EPA and DHA supplementation
Dietary Supplement: Placebo — Subjects will be given 3g/d of soy oil - 5 capsules per day.
  Arms: Placebo

SUMMARY:
It has been demonstrated that EPA and DHA supplementation may have anti-inflammatory properties in several chronic diseases, namely, diabetes, obesity, and in rheumatoid arthritis, although not with controversy. Systemic lupus erythematosus (SLE) and Antiphospholipid Antibody Syndrome (AAS) are autoimmune diseases characterized by a chronic inflammatory state which is associated with the disease´s clinical symptoms. Thus, we hypothesized that EPA and DHA supplementation may beneficially affect the inflammatory cytokine profile and clinical features of LES and AAS patients.

ELIGIBILITY:
Inclusion Criteria:

• Age between 7 and 40 years

Exclusion Criteria:

* Cardiovascular dysfunction
* Rhythm and conduction disorders
* Musculoskeletal disturbances
* Kidney and pulmonary involvements
* Peripheral neuropathy
* Use of tobacco
* Treatment with lipid-lowering or hypoglycemic drugs
* Fibromyalgia
* Use of chronotropic or antihypertensive drugs
* Physically active subjects

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cytokine profile (serum levels of IL-1B, IL-2, IL-4, IL-6, IL-8, IL-10, TNF-alpha, IFN-y) | 4 months
  Cytokines´ serum levels (pg/ml) will be assessed by Elisa kits.
Endothelial function | 4 months
  Endothelial function assessed by flow mediated dilatation (FMD).

SECONDARY OUTCOMES:
Clical features | 4 months
  Disease activity - assessed by SLEDAI score
Clinical features | 4 months
  Quality of life - assessed by SF-36 questionaire
Clinical features | 4 months
  Fatigue - assessed by 2 questionaires - Chalders´Fatigue Scale and Fatigue Severity Scale (FSS)
Clinical features | 4 months
  Body composition - lean (Kg) and fat mass (Kg) assessed by air displacement pletysmography (BOD POD).

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital - University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Felau SM, Sales LP, Solis MY, Hayashi AP, Roschel H, Sa-Pinto AL, Andrade DCO, Katayama KY, Irigoyen MC, Consolim-Colombo F, Bonfa E, Gualano B, Benatti FB. Omega-3 Fatty Acid Supplementation Improves Endothelial Function in Primary Antiphospholipid Syndrome: A Small-Scale Randomized Double-Blind Placebo-Controlled Trial. Front Immunol. 2018 Mar 2;9:336. doi: 10.3389/fimmu.2018.00336. eCollection 2018. PMID 29552010